CLINICAL TRIAL: NCT02563366
Title: Effect of Bone Marrow-derived Mesenchymal Stem Cells (BM-MSCs) on Recovery of Poor Early Graft Function Post Kidney Transplantation From Chinese Donation After Citizen Death (DCD): A Multi-center Randomized Controlled Trial
Brief Title: Effect of BM-MSCs on Early Graft Function Recovery After DCD Kidney Transplant.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Changxi Wang, Director of Organ Transplant Center, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSCs-KTx-DCD-150925
Record Dates: First submitted 2015-09-26; First posted 2015-09-30 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Kidney Transplantation; Acute Kidney Tubular Necrosis
Keywords: kidney transplantation; mesenchymal stem cell therapy; poor early graft function; delayed graft function; ischemia reperfusion injury; donation after cardiac death
MeSH Terms: conditions — Kidney Tubular Necrosis, Acute; Delayed Graft Function; Reperfusion Injury | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- MSCs group (Experimental): Patients with early poor graft function receive allogeneic BM-MSCs at the dose of 1*10^6/kg every week for four consecutive doses.
  Interventions: Other: BM-MSCs
- Control group (Placebo Comparator): Patients with early poor graft function receive placebo of MSCs, i.e. saline every week for four consecutive doses.
  Interventions: Other: Saline

INTERVENTIONS:
Other: BM-MSCs — BM-MSCs are from third-party healthy volunteer donors.
  Other Names: allogeneic bone marrow-derived MSCs
  Arms: MSCs group
Other: Saline — Saline is the placebo of MSCs in this study.
  Arms: Control group

SUMMARY:
This study is designed to investigate whether allogeneic bone marrow-derived mesenchymal stem cells (BM-MSCs) can promote function recovery in patients with poor early graft function after kidney transplantation from Chinese Donation after Citizen Death (DCD). DCD kidney transplant recipients with poor early graft function (with or without dialysis) post transplant are equally randomized into MSCs group or control group. Patients in MSCs group are administered MSCs treatment. Allogeneic BM-MSCs (1*10^6/kg) from third party are given intravenously for four consecutive doses every week after enrollment. Patients in control group receive placebo. Renal allograft function (eGFR), rejection, patient/graft survival and severe adverse events up to 12 months post enrollment are monitored.

ELIGIBILITY:
Inclusion Criteria:

* Primary kidney transplantation
* Kidneys are from donation after Chinese citizen death
* Poor early graft function with or without dialysis after transplantation
* Patient is willing and capable of giving written informed consent for study participation and able to participate in the study for 12 months

Exclusion Criteria:

* Secondary kidney transplantation
* Combined or multi-organ transplantation
* Women who are pregnant, intend to become pregnant in the next 1 years, breastfeeding, or have a positive pregnancy test on enrollment or prior to study medication administration
* Panel reactive antibody (PRA)>20% or CDC crossmatch is positive
* Donors or recipients are known hepatitis C antibody-positive or polymerase chain reaction (PCR) positive for hepatitis C
* Donors or recipients are known hepatitis B surface antigen-positive or PCR positive for hepatitis B
* Donors or recipients are known human immunodeficiency virus (HIV) infection
* Patients with active infection
* Recipients with a history of substance abuse (drugs or alcohol) within the past 6 months, or psychotic disorders that are not capable with adequate study follow- up.
* Patients with severe cardiovascular dysfunction
* WBC<3*10^9/L or RBC <5g/dL
* Highly allergic constitution or having severe history of allergies.
* Patients with active peptic ulcer disease, chronic diarrhea, or gastrointestinal problem affect absorption
* Patients with a history of cancer within the last 5 years
* Prisoner or patients compulsorily detained (involuntarily incarcerated) for treatment or either a psychiatric or physical (e.g. infectious disease) illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate | 1 month
  eGFR at one month post transplant

SECONDARY OUTCOMES:
Estimated glomerular filtration rate | 12 months
  eGFR up to 12 months post transplant
Proportion of normal renal function recovery | 12 months
Time to renal function recovery (days) | 12 months
acute rejection rate | 12 months
  Acute rejection rate according to Banff 2013 criteria up to 12 months post transplant
patient and graft survival rate | 12 months
  patient and graft survival rate up to 12 months post transplantation
Incidence of severe adverse events | 12 months
  Incidence of severe adverse events up to 12 months post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Changxi Wang, M.D., Ph.D, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Peng Y, Ke M, Xu L, Liu L, Chen X, Xia W, Li X, Chen Z, Ma J, Liao D, Li G, Fang J, Pan G, Xiang AP. Donor-derived mesenchymal stem cells combined with low-dose tacrolimus prevent acute rejection after renal transplantation: a clinical pilot study. Transplantation. 2013 Jan 15;95(1):161-8. doi: 10.1097/TP.0b013e3182754c53. PMID 23263506
- See also: Previous publication — http://www.ncbi.nlm.nih.gov/pubmed/23263506